CLINICAL TRIAL: NCT00718627
Title: Open, Prospective, Uncontrolled, Multicentre Study to Evaluate The Safety and Efficacy of Multiple Applications of Liver Cell Suspension Into The Portal Vein in Children With Urea Cycle Disorders (UCDs)
Brief Title: Human Heterologous Liver Cells for Infusion in Children With Urea Cycle Disorders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cytonet GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCD02; CCD02 (Other: cytonet); 2006-000136-27 (EudraCT Number)
Record Dates: First submitted 2008-07-16; First posted 2008-07-18 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-02

CONDITIONS: Urea Cycle Disorders; Carbamoylphosphate Synthetase I Deficiency; Ornithine Transcarbamylase Deficiency; Citrullinemia
Keywords: Urea cycle Disorders; Carbamoylphosphate synthetase I deficiency; Ornithine transcarbamoylase deficiency; Argininosuccinate synthase deficiency; Citrullinemia; newborns; infants; liver cell transplantation; liver cell infusion
MeSH Terms: conditions — Urea Cycle Disorders, Inborn; Ornithine Carbamoyltransferase Deficiency Disease; Citrullinemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HHLivC Therapy Group (Experimental)
  Interventions: Biological: Human Heterologous Liver Cells

INTERVENTIONS:
Biological: Human Heterologous Liver Cells — Multiple applications of liver cell suspension for infusion

SUMMARY:
Urea cycle disorders are rare inherited diseases that generally have a poor outcome. In this study, neonates and infants with UCD will be included within the first 3 months of life and will be treated by repetitive application of human liver cells to reduce the risk of neurological deterioration while awaiting OLT.

DETAILED DESCRIPTION:
Urea cycle disorders are rare inherited diseases that generally have a poor outcome, especially with onset of the disease in the neonatal period. UCDs are caused by a deficiency of one of six enzymes responsible for removing ammonia from the bloodstream. Instead of being converted into urea which is removed from the body with the urine, ammonia accumulates in UCD patients leading to brain damage or death. In the light of a mortality rate of > 50% at the age of 10 years the current pharmacological and dietary therapy is of modest success. Furthermore, mental retardation, cerebral palsy and other neurological sequelae are common among surviving patients.

In the last years, orthotopic liver transplantation (OLT) has become the best therapeutic option for UCD with long-term survival rates of about 90%. However, in the first weeks of life OLT still is technically demanding and prone to complications. With larger size of the recipient, the technical problems with OLT decrease considerably. The increased body weight usually achieved at the age of more than 8 weeks is related to a major reduction in transplantation related morbidity. Stabilization of metabolism until the patient can undergo OLT is essential.

In this study, neonates and infants with UCD will be included within the first 3 months of life and will be treated by repetitive application of human liver cells. In the last consequence, the aim of this new therapy option is to supply a sufficient amount of healthy liver cells to compensate for the metabolic defect and to reduce the risk of neurological deterioration while awaiting OLT.

ELIGIBILITY:
Inclusion Criteria

* Neonates and infants up to the age of ≤ 3 months with prenatally or postnatally confirmed urea cycle disorder and
* Children aged > 3 months up to ≤ 5 years of age with unstable metabolism and confirmed urea cycle disorder of either:

  * Carbamylphosphate synthetase I [CPSD] or
  * Ornithine transcarbamylase [OTCD] or
  * Argininosuccinate synthetase [Citrullinaemia]
* A DNA analysis will further confirm diagnosis prior to or after inclusion according to the protocol.

  * Accessibility of the portal vein
  * Plasma ammonia level ≤ 250 μmol/l
  * Written informed consent

Exclusion Criteria

* Structural liver disease (cirrhosis, portal hypertension), or venoocclusive diseases
* Portal vein thrombosis
* Body Weight ≤3.5 kg
* Carrier of the human immuno-deficiency virus (HIV)
* Any other contraindication for immunosuppression
* Presence of acute infection at the time of inclusion
* Participation in other clinical trials or received experimental medication within the last 30 days
* Live vaccination planned during the course of the study
* Live vaccination within 4 weeks prior to beginning of study
* Allergic disposition against contrast medium used in study and/or antibiotics used in the manufacturing process
* Required valproate therapy
* Severe coagulopathy or thrombocytopenia
* Known diagnosis of hereditary thrombophilia (e.g. Factor V Leiden, Prothrombin 20210A variant) or parental history of hereditary thrombophilia and absense of thrombophilia testing in subject
* Cancer, severe systemic or chronic disease other than study indication (urea cycle deficiency)

Ages: 1 Day to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2008-07; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Safety of the application of liver cells, safety of the placement of an application catheter to the portal vein. | 7 - 15 weeks

SECONDARY OUTCOMES:
Changes in 13C urea formation. Changes in the respective enzyme activity in liver biopsies from the explanted organ compared to the enzyme activity in the liver before cell application. | 7-15 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Georg Hoffmann, Prof., Principal Investigator — University Children's Hospital
Locations (2):
- Germany (2):
  - University Children's Hospital, Heinrich-Heine University, Düsseldorf
  - University Children's Hospital, Heidelberg